CLINICAL TRIAL: NCT01142518
Title: A Prospective Analysis of MS Patients After Starting or Restarting Baseline Treatment With Interferon Beta 1a After the Use of Escalation Treatment
Brief Title: An Observational Study of Multiple Sclerosis (MS) Patients Starting or Restarting Baseline Treatment With Interferon Beta 1a After the Use of Escalation Treatment With Mitoxantrone
Acronym: RETURN
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Norbert Zessack/Head of Medicine BU Neurology, Merck Serono GmbH Germany, an affiliate of MerckKGaA, Darmstadt, Germany
Other Study IDs: IMP28169
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Interferon beta-1a; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples

INTERVENTIONS:
Drug: Interferon beta 1a — Interferon beta 1a was administered at a dose of 44 μg x 3 as a subcutaneous self-injection.
  Other Names: Rebif®

SUMMARY:
This was an open-label, multicentric, prospective, post-marketing surveillance (PMS) study to investigate whether baseline treatment with high-dose interferon beta 1a (Rebif 44 μg x 3 ), administered at a high frequency, leads to maintenance of stabilisation of the course of the disease in MS subjects previously treated with mitoxantrone. The previous mitoxantrone treatment of the included MS subjects was conducted in the course of a so-called escalation according to the immunomodulatory escalation treatment plan. An additional important aspect of the problem was the collection of safety and tolerance data during the observation phase.

DETAILED DESCRIPTION:
The treatment of relapsing-remitting MS with interferon-beta has established itself as first-choice treatment. In previous clinical studies, the interferon-beta 1a (Rebif) used within the scope of this PMS study has demonstrated significant efficacy in all aspects of treatment - magnetic resonance imaging (MRI) data, relapse rate, progression of disability of MS. The PRISMS-4 study demonstrated that treatment with Rebif reduces the frequency and severity of clinical relapses over 4 years and slows the progression of disability.

In the course of treatment escalation according to the Multiple Sklerose Therapie Konsensus Gruppe (MSTKG) guidelines, MS subjects with correspondingly high disease activity were predominantly put on mitoxantrone. The duration of treatment is on principle limited by a cumulative lifelong total dose of 140 mg/m2 body surface area, which may not be exceeded due to the known cardiologic adverse effects. If the cumulative mitoxantrone maximum dose is reached and if the subject is in a stable condition, the question of further treatment options presents itself. One possibility is the so-called 'deescalation', that is, the return to immunomodulating baseline treatment.

Currently there is an increasing number of subjects who are in this phase of the disease and are eligible for corresponding treatment decisions.

OBJECTIVES

Primary objective:

* To systematically investigate the safety, benefit and course of Rebif (44 μg x 3 ),treatment in a larger number of subjects and to subject these data to standardized analysis

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinically demonstrated diagnosis of MS and present relapses
* Subjects who were relapse-free for the past 6 months with an Expanded Disability Status Scale (EDSS) range between 2 and 6
* Subjects who had a stable disease status during the past few months
* The last administration of mitoxantrone had been more than 3 months previously. In addition, the mitoxantrone treatment was given for at least a 12-month period, but for not more than 24 months, within a total dosage of 60-120 mg/m2 body surface area

Exclusion Criteria:

* Subjects with MS with secondary progression (SPMS) without relapse activity, pregnant or breast-feeding patients, as well as subjects with contraindications
* Subjects with existing systemic concomitant diseases (e.g. diabetes, heart, liver or kidney diseases)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A group of MS subjects who will be treated with Rebif after being previously treated with mitoxantrone
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2005-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Stabilization of the course of the disease in MS subjects previously treated with mitoxantrone | 24 months

SECONDARY OUTCOMES:
Safety and tolerance of the treatment | 24 months
  Assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Norbert Zessack, Study Director — Merck Serono GmbH, Germany